CLINICAL TRIAL: NCT07194239
Title: Life-Style Medicine for Chronic Musculoskeletal Pain in Older People: A Pragmatic, Randomized Controlled Clinical Trial
Brief Title: Life-Style Medicine for Chronic Musculoskeletal Pain in Older People
Acronym: lifestyle med
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Regina Wing Shan Sit, Associate Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025.553; 2025.553 (Other: Hospital Authority Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-17; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Musculoskeletal; Pain Management; Chronic Pain; Musculoskeletal Pain
Keywords: Musculoskeletal pain; lifestyle medicine; older people; health coaching; Chronic Musculoskeletal Pain; Behavior change
MeSH Terms: conditions — Agnosia; Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (No Intervention): Patients allocated to the Waitlist arm will continue receiving their "usual care" without any additional intervention until they have completed the outcome assessment at 24 weeks.
- Intervention group (Experimental): A coaching context to enhance the well-being of individuals and to facilitate the achievement of their health-related goals. The coach will negotiate and set personalized health goals with participants, ensuring the goals are realistic, achievable, and aligned with their needs.
  Interventions: Behavioral: Lifestyle medicine Health coaching

INTERVENTIONS:
Behavioral: Lifestyle medicine Health coaching — Participants assigned to this group will have 4 face-to-face sessions with the health coach. Lifestyle modifications with the aim of pain reduction will be determined in a shared decision-making approach. Lifestyle modifications will be based on the 6 pillars of lifestyle medicine: Physical activity, Healthy eating, Stress reduction, Sleep restoration, Social Support, and Avoiding risky substances. The health coach will make use of motivational techniques such as motivational interviewing to guide and assist participants in realizing the lifestyle modifications.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to determine the clinical effectiveness of lifestyle medicine in reducing chronic musculoskeletal pain in older adults, as measured by pain intensity, pain interference, self-management efficacy, stress level, sleep quality, healthier diet, better quality of life, and cost-effectiveness, compared to a waitlist control group.

Participants will be randomly assigned to either the intervention or the waitlist group. The intervention group will meet the health coach face-to-face for four sessions to negotiate and set personalized health goals. The waitlist control group will continue to receive usual care without any additional intervention for 24 weeks. Both groups will complete three assessments: at the start of the study, one month after the intervention, and three months after the intervention. The waitlist control group will be offered the same intervention after completing the study.

ELIGIBILITY:
Inclusion Criteria:

* chronic musculoskeletal pain, defined as pain that lasted for more than 3 months persistently or intermittently, including regional pain (joints, limbs, back, and/or neck)
* a degenerative joint condition, such as osteoarthritis, and/or musculoskeletal complaints that fall under the classification of the International Classification of Disease-11 as "chronic primary musculoskeletal pain" or "chronic secondary musculoskeletal pain"
* Pain intensity score ≥ 4 on a numerical rating scale of 10
* stable baseline physical activity
* ability to understand written and verbal Chinese

Exclusion Criteria:

* patient with cancer-related pain
* inflammatory rheumatic disease
* a recent history of stroke or major surgery in the past 6 months
* terminal illness
* serious mental illness
* severe or uncontrolled heart disease
* comorbid conditions that might impede active participation in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Severity score | Week 0, 12, 24
  The Brief Pain Inventory (BPI) is a self-report questionnaire that assesses the intensity of pain and its effects on daily functioning. BPI- Severity measures the intensity of pain. Participants are asked to rate their pain on a 0-10 Numeric Rating Scale for their pain experienced at its "worst," "least," "average," and "now" over the past 24 hours. Higher scores indicate greater pain severity.

SECONDARY OUTCOMES:
BPI-Interference | week 0, 12, 24
  The Brief Pain Inventory (BPI) is a self-report questionnaire that assesses the intensity of pain and its effects on daily functioning. BPI- Interference measures the level of interference as a result of pain. Participants are asked to rate the level of interference experienced over the past 24 hours on a 0-10 Numeric Rating Scale for seven interference items: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Higher scores indicate greater pain interference.
Pain-Self Efficacy questionnaire | Week 0 12, 24
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item self-report questionnaire that measures an individual's confidence in performing daily activities and managing life despite experiencing persistent pain. Each item is measured on a 7-point Likert scale (ranging from 0 to 6). The items assess confidence in performing tasks such as household chores, socializing, working, and coping without medication. A higher total score indicates a stronger belief in managing pain effectively.
Chinese International Physical Activity Questionnaire (Short form) | Week 0, 12, 24
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) is an 8-item self-report questionnaire designed to assess the overall physical activity over the past 7 days. Questionnaire items measure the frequency (days) and duration (time) of activities, including walking, moderate-intensity, vigorous-intensity activities, and sedentary behavior.
Chinese Short Food Frequency Questionnaire | Week 0, 12, 24
  The Food Frequency Questionnaire (FFQ) consists of 50 food items reflecting the typical dietary intake of Chinese older adults in Hong Kong. The FFQ captures habitual food consumption by combining frequency and portion data to quantify nutrient and food group intake. Participants report the frequency of consumption and portion size for each item, allowing estimation of average daily intake.
10-item Perceived Stress Scale (PSS-10) | Week 0, 12, 24
  The 10-item Perceived Stress Scale (PSS-10) is a self-reported questionnaire that measures the degree to which individuals perceive their lives as unpredictable, uncontrollable, and overloaded over the past month. The items are rated on a 5-point Likert scale from "never" to "very often". Items include six negatively phrased items assessing perceived helplessness and four positively phrased items measuring perceived self-efficacy or coping. Scores for the positively worded items are reverse-coded, and the total score ranges from 10 to 50, with higher scores indicating greater perceived stress.
7-item Insomnia Severity Index (ISI) | Week 0, 12, 24
  The 7-item Insomnia Severity Index (ISI) is a self-report questionnaire that assesses the severity and impact of insomnia symptoms. It evaluates difficulties with sleep onset, sleep maintenance, early morning awakening, satisfaction with current sleep patterns, interference with daily functioning, the degree to which the sleep problem is noticeable to others, and the level of distress caused by the sleep problem. Each item is rated on a 5-point scale, ranging from 0 (no problem) to 4 (very severe problem), with total scores ranging from 0 to 28. Higher scores indicate more severe insomnia.
Lubben Social Network Scale-6 (LSNS-6) | Week 0, 12, 24
  The Lubben Social Network Scale-6 (LSNS-6) is a brief, 6-item self-report questionnaire designed to assess social engagement and the size of social networks among older adults by measuring perceived social support from family and friends. Items include questions on relatives and friends seen or heard from at least once a month, and those the respondent feels comfortable talking to or can call on for help. Scores range from 0 to 30, with higher scores indicating stronger social networks and lower risk of social isolation.
EuroQuol-5D-5L (EQ-5D-5L) | Week 0, 12, 24
  The EuroQuol-5D-5L (EQ-5D-5L) assesses health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels, ranging from "no problems" to "extreme problems". The questionnaire also includes a visual analogue scale (VAS) for rating overall health on a scale from 0 (worst) to 100 (best).
Quantity of smoking and alcohol consumption | Week 0, 12, 24
  The participant's past or current history of smoking and the level of alcohol consumption over the past year will be recorded.
Quality-adjusted life years (QALYs) on EQ-5D-5L | Week 0, 12, 24
  Quality-Adjusted Life Years (QALYs) based on the EQ-5D-5L are calculated by multiplying a health utility value, which ranges from 0 (equivalent to death) to 1 (perfect health), by the time spent in that health state. These utility values are derived from the EQ-5D-5L questionnaire responses using country-specific value sets that reflect societal preferences for different health conditions. This calculation provides a combined measure of both the quality and length of life, commonly used to evaluate the effectiveness and cost-efficiency of healthcare interventions.